CLINICAL TRIAL: NCT06709859
Title: A Phase II Trial to Evaluate the Efficacy and Safety of Afatinib Combined With Chemotherapy as Conversion Therapy in Unresectable EGFR Sensitive Mutation-positive Stage III Non-small Cell Lung Cancer
Brief Title: Afatinib Combined With Chemotherapy as Conversion Therapy in Unresectable EGFR Sensitive Mutation-positive Stage III NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Public Health Clinical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWLCZXEC2024-56-2
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Conversion Therapy; Afatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Afatinib plus chemotherapy (Experimental): Patients with unresectable EGFR sensitive mutation-positive stage III NSCLC will receive 3-4 cycles of afatinib plus chemotherapy as the conversion treatment (afatinib 40mg qd; carboplatin (AUC 5) on day 1, and pemetrexed (500 mg/m2 for non-squamous carcinoma) or nab-paclitaxel (260 mg/m2 for squamous carcinoma) d1 q3w), and then surgery will be provided for patients who are suitable for primary tumor resection. Maintenance treatment with afatinib 40mg qd will continue up to 2 years or disease progression after surgery.
  Interventions: Drug: Afatinib plus chemotherapy as conversion treatment

INTERVENTIONS:
Drug: Afatinib plus chemotherapy as conversion treatment — Patients with unresectable EGFR sensitive mutation-positive stage III NSCLC will receive 3-4 cycles of afatinib plus chemotherapy as the conversion treatment, and then surgery will be provided for patients who are suitable for primary tumor resection.

SUMMARY:
This is a phase II, single-arm study to evaluate the efficacy and safety of Afatinib plus chemotherapy as conversion treatment in patients with unresectable EGFR sensitive mutation-positive stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
This single-arm, open-label, prospective phase II clinical trial was designed to evaluate the efficacy and safety of afatinib plus chemotherapy as conversion treatment in patients with unresectable EGFR sensitive mutation-positive stage III non-small cell lung cancer.

The primary endpoint was the rate of NSCLC converting to resectable tumors. The secondary endpoints included R0 resection rate, major pathological response (MPR) rate, pathological complete response (pCR) rate, tumor downstaging rate, objective response rate (ORR), disease control rate (DCR), 1-year event-free survival (EFS) rate, EFS and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed diagnosis of unresectable Stage III non-small cell lung cancer as judged by the investigator.
* Tissue or blood samples tested and confirmed to be positive for EGFR sensitive mutation
* ECOG Performance Status of 0-1
* At least one measurable lesion according to RECIST 1.1
* Adequate organ and marrow function

Exclusion Criteria:

* Histologically or cytologically confirmed combined SCLC and NSCLC, large cell neuroendocrine carcinoma, and sarcoma-like carcinoma
* The presence of malignant pleural effusion
* Prior systemic anti-cancer therapy for non-small cell lung cancer
* Prior local radiotherapy for NSCLC
* Patients with uncontrolled gastrointestinal diseases that may affect the absorption of test drugs (such as Crohn's disease, ulcerative colitis, absorption disorders, or diarrhea of any cause ≥ Grade 2 CTCAE) according to the investigator's assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of NSCLC converting to resectable tumors | Up to 12 weeks
  The proportion of unresectable NSCLC patients who are converted to being suitable for surgery after 3-4 cycles afatinib plus chemotherapy.

SECONDARY OUTCOMES:
R0 resection rate | immediately after the surgery
  The proportion of R0 resection in patients who receive surgery
Major pathologic response (MPR) Rate | Up to 12 weeks
  The proportion of patients who achieve MRP among those receiving surgery
Pathologic complete response (pCR) Rate | Up to 12 weeks
  The proportion of patients who achieve pCR among those receiving surgery
Tumor downstaging rate | Up to 12 weeks
  The proportion of patients who reach the successful downstaging criteria for NSCLC
Objective response rate (ORR) | Up to five years
  The proportion of patients who have a complete response (CR) or partial response (PR).
Disease control rate (DCR) | Up to five years
  The proportion of patients who have a best overall response of CR, PR, or stable disease (SD).
Event-free survival (EFS) | Up to five years
  The length of time after initial administration the patient remains free of recurrence/progression or death, whatever the cause.
The 2-year progression-free survival (PFS) rate | Up to two years
  The proportion of patients who are event-free.
Overall Survival (OS) | Up to five years
  The length of time after initial administration the patient remains alive

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhang, PhD, Principal Investigator — Shandong Public Health Clinical Center
Locations (1):
- Shandong Public Health Clinical Center, Jinan, Shangdong, China

IPD SHARING:
Plan to Share IPD: No